CLINICAL TRIAL: NCT02568007
Title: Effects of Cyproheptadine on Growth and Behavior in Pediatric Feeding Disorders
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to enroll adequate participants
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Praveen Goday, Professor of Pediatric Gastroenterology, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 798217
Record Dates: First submitted 2015-09-03; First posted 2015-10-05 (Estimated); Results first posted 2020-01-31 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Feeding Behaviors
MeSH Terms: conditions — Feeding Behavior | interventions — Cyproheptadine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- No Cyproheptadine treatment (No Intervention): Patients will receive standard of care behavior and nutritional interventions. They will not receive cyproheptadine.
- Continuous Cyproheptadine (Experimental): Patients will receive standard of care behavior and nutritional interventions. They will receive cyproheptadine every day for a total of two months. Standard dose of 0.25 mg/kg divided BID will be used.
  Interventions: Drug: Cyproheptadine
- Cycled Cyproheptadine (Experimental): Patients will receive standard of care behavior and nutritional interventions. They will receive cyproheptadine every day for two weeks cycled with no cyproheptadine given for two weeks for a total of two months. Patients on cycled dosing will be given cyproheptadine for two weeks, then no medication for two weeks; repeating this cycle for the two month duration of study
  Interventions: Drug: Cyproheptadine

INTERVENTIONS:
Drug: Cyproheptadine
  Arms: Continuous Cyproheptadine; Cycled Cyproheptadine

SUMMARY:
The purpose of this study is to examine the effect of standard dosing of cyproheptadine for both cycled and continuous administration, as compared to no medication, on appetite stimulation and growth in the pediatric gastroenterology feeding team patient population. The secondary aim is to evaluate the effect, if any, of the suspected tachyphylaxis that is commonly associated with cyproheptadine use. The third aim will be to examine the type and duration of side effects of cyproheptadine in this population. The ultimate goal will be to create a standardized protocol for cyproheptadine therapy in children with feeding disorders and suboptimal growth.

DETAILED DESCRIPTION:
BACKGROUND, SIGNIFICANCE, AND RATIONALE Failure to thrive or inadequate weight gain is a frequent complaint amongst patients seen by general pediatricians and pediatric gastroenterologists. The reasons behind this diagnosis vary widely including, but not limited to feeding disorders of diverse etiologies, poor environmental structure and inadequate intake, medication side effects, swallowing disorders, and a variety of underlying organic diseases. For most feeding disorders, behavioral feeding techniques and strategies to increase caloric intake is utilized to correct the suboptimal growth. However, feeding disorders are sometimes so imprinted that behavioral interventions may be insufficient to promote ideal growth or, if sufficient for growth, are inadequate in helping children avoid or graduate from nutritional support such as enteral tubes. For this reason, medications that promote and stimulate appetite and weight gain are frequently used in children with feeding disorders.

In pediatric gastroenterology practice, cyproheptadine is the most commonly used drug for appetite stimulation, weight gain, and feeding intolerance in younger children with feeding disorders. A first generation histamine and serotonin antagonist, cyproheptadine is thought to promote appetite stimulation and weight gain by increasing insulin-like growth factor-1 (IGF-1) concentration. It may also interact with receptors in the ventromedial hypothalamus and exert hormonal effects. While the exact mechanism of action is still being investigated, several studies have evaluated the benefits of cyproheptadine in select patient groups, including patients with cystic fibrosis, cancer, undernourished children, and children with feeding disorders. These studies have all reported that cyproheptadine promotes weight gain and stimulates appetite. Reported side effects of cyproheptadine in these studies are primarily related to drowsiness which tends to significantly improve or resolve within two weeks of use. Another undesired effect is the development of drug tolerance, i.e. tachyphylaxis. To avoid this, it is common clinical practice to cycle on and off the medication a few weeks each month.

While a few studies report outcomes of the use of cyproheptadine in children with feeding disorders or failure to thrive, these studies have enrolled only small patient cohorts and there are no randomized trials in children enrolled in a feeding team program. Two recent studies examined the role of cyproheptadine in patients who are undernourished or followed in pediatric feeding programs. However, a randomized study examining the effects of continuous cyproheptadine versus a fixed cycled medication dosing versus abstaining from medication has not been performed in the pediatric gastroenterology population.

OUTCOME MEASURES:

Number of Participants in Study: The total number of patients required for this study is 75 (25 in each group). The groups consist of three treatment arms:

1. continuous use of cyproheptadine
2. cycled cyproheptadine or
3. no drug intervention

This number was derived from looking at past statistical data from other studies and using similar power, alpha error, and beta error. Investigators used Analysis of Variance (ANOVA) analysis for multiple groups looking at repeat measures within factors. Alpha error was 0.05, Power 0.95.

Data Collection: The following categories of data will be collected (see subsections list below): medical record number (MRN), demographics, feeding behavior, side effects experience from use cyproheptadine, 24 hour diet recalls, medical history, and anthropometrics.

Demographic Information: Data will be collected as part of the demographics questionnaire. This includes participant's age, sex, ethnicity, identification of primary caretaker, caretaker's relation to participant, caretaker education level, and caretaker marital status.

Feeding Behavior Questionnaire: Patients/parents will complete the Mealtime Behavior Questionnaire (MBQ). Participants' guardians will complete the Mealtime Behavior Questionnaire (MBQ). This is a validated, 31-item, parent-report questionnaire assessing the mealtime behavior structure in young children above 2 years.

The questionnaire measures variables including:

1. food refusals/avoidance
2. food manipulation
3. mealtime aggression and
4. choking/gagging/vomiting related to meals.

Each behavior is assigned a frequency scale with 1 corresponding to "never" and 5 corresponding to "always." The MBQ then consist of a total score and four subcategory scores (listed above).

24 Hour Diet Recall: Guardians of participants will be questioned weekly regarding oral intake (type of food consumed and amount) over the past 24 hrs. Caloric intake will be calculated based on these recalls and compared across duration of study.

Cyproheptadine Side Effect Questionnaire: Guardians will undergo weekly questionnaire looking at common side effects of cyproheptadine. A list of side effects will be read to the participant's guardians with positive (yes) or negative (no) replies if the participant has experienced individual side effects since the last survey.

Medical Information: Data collected will include anthropometrics at initial and final visit (weight, height, BMI, mid-arm circumference, upper arm skin fold), current and past medical diagnoses and surgeries, current medications, current gastrointestinal symptoms, dependence on tube feeds

RISK CATEGORY:

Research not involving greater than minimal risk to the children.

KNOWN SIDE EFFECTS OF CYPROHEPTADINE:

Cyproheptadine has both antihistamine and antiserotonergic and has side effects related to these mechanisms. These side effects include drowsiness or sleepiness, confusion, excitement, fatigue, insomnia, hallucinations, blurred vision, tinnitus, dizziness, tachycardia, increase perspiration, appetite stimulation, weight gain, constipation, diarrhea, changes in frequency of urination, thickening of secretions, and dry mucus membranes. Over-dosage can results in atropine-like effects as well as central nervous depression, convulsions.

SECURITY OF DATA COLLECTED:

All investigators have received Health Insurance Portability and Accountability Act (HIPAA) training and a certificate of completion for the Collaborative Institutional Training Initiative (CITI) training course on the protection of human research subjects before starting the review. Information derived from questionnaires, data collection will be compiled on one central data collection form. These forms will be coded (have a special identifier number that is linked to patient's MRN). The central database used for data collection will be password protected. A separate secure (password protected) database will link the coding number to the patient's MRN. Only the principal investigator (PI), co-investigators and the members of the study team will be gathering the data and have access to the study database. Paper records will be locked in file cabinets within the Gastroenterology office area and electronic records will be stored in password-protected computers. Each subject's identifying number and related electronic data will be kept on a secured, password-protected database that provides access only to the PI and research staff. Only authorized research personnel will have access to the databases and paper records.

PROVISION FOR THE PROTECTION OF PRIVACY OF SUBJECTS (confidentiality, health and financial risks) AND TO MAINTAIN THE CONFIDENTIALITY OF DATA:

Data will be stored on Medical College of Wisconsin secured shared drives.

PROVISIONS FOR MONITORING DATA TO ENSURE THE SAFETY OF SUBJECTS; AND ADDITIONAL SAFEGUARDS TO PROTECT THE RIGHTS AND WELFARE OF SUBJECTS WHO ARE LIKELY TO BE VULNERABLE:

The PI will monitor the health of all patients in the study per standard clinical practice. Primary and Co-investigators will monitor protocol adherence and supervise data collection, entry, and analysis.

ANTICIPATED BENEFITS ASSOCIATED WITH THE PROTOCOL (value or desired outcome / advantage) TO HUMAN RESEARCH PARTICIPANTS AND SOCIETY (medical, psychosocial, altruistic) Anticipated direct benefits of this study include the improvement in appetite/behavior and growth amongst the patients receiving cyproheptadine. These benefits may also be present in group abstaining from cyproheptadine due to standard education that is given to all groups. However, the investigators anticipate these benefits to be significantly lower in this group as compared to patients who are on cyproheptadine. Long-term benefits include the creation and utilization of a protocol outlining the use of cyproheptadine in feeding team patients. The results of this study will also address the side effect profile of cyproheptadine in this population. It may also further investigators' knowledge of the treatment approaches that are most successful, allowing physicians to develop standardized care to better serve these patients and their families.

STOPPING POINTS THAT WOULD NOT ALLOW THE STUDY TO CONTINUE AS PROPOSED:

Stopping points for the study include achieving adequate information on enough of the goal subjects, inability to obtain enough data, or patients/caregivers electing to discontinue the study.

DESCRIBE HOW THE CONSENT (AND ASSENT, IF APPLICABLE) PROCESS WILL TAKE PLACE. INCLUDE A LIST OF APPROPRIATELY TRAINED PERSONNEL WHO WILL BE INVOLVED.

Written informed consent for participation will be obtained from guardians for their child's participation. Consent will be obtained by study personnel at the participant's appointment in the GI Clinic. Participants' consent will allow for accessing information collected for program evaluation/clinical purposes. Participants' guardians will have the option of having the consent document read aloud to them to facilitate understanding. Copies of signed consent documents will be given to participants' guardians. Consent will be obtained by the study's principal investigator, co-investigators, or members of the research team. As additional research staff or team members are added, their names will be submitted to the International Review Board (IRB) as a protocol amendment to allow them to obtain consent.

PROCEDURES TO BE EMPLOYED IN ANALYZING DATA (including a power analysis) AND THE ANTICIPATED SIGNIFICANCE OF THE PROPOSED STUDY Analyses will be conducted with Statistical Package for the Social Sciences (SPSS) and Statistical Analysis System (SAS) software programs. Probability levels of < .05 will be used as cut offs for statistical significance. Descriptive analyses will examine distribution normality and the extent to which parametric test assumptions are met. Descriptive analyses will also provide summary information about participant characteristics. Pearson correlations will be used to examine relationships between continuous variables, while chi square analyses will examine associations between categorical variables.

The key significance of this study is the analysis of the effect that cyproheptadine has on stimulating weight gain and improving behaviors associated with feeding. In addition, it will help give clear comparison between the use of continuous versus cycled cyproheptadine. Cyproheptadine has been suspected to have tachyphylaxis after a couple weeks and many practitioners implement cycling of medication without clear evidence supporting this practice. Investigators expect after this study to be able to design a protocol regarding use of cyproheptadine in feeding team patients.

FINANCIAL RELATIONSHIPS:

There are no financial relationships or interests to disclose.

ADVERTISEMENTS / FLIERS (how will they be used / distributed):

None will be used

ELIGIBILITY:
Inclusion Criteria:

* All children aged 1-10 years, presenting to initial intake appointment with the Pediatric Gastroenterology Feeding Team Clinic at the Children's Hospital of Wisconsin (CHW), with BMI Z score of < or equal to 0 (normal WHO BMI defined as Z score of -1 to 1), who have a parent willing to participate, will qualify for inclusion in the study. Children with vomiting due to presumed volume intolerance may be included in the study.

Exclusion Criteria:

* Untreated organic disease Anatomical barrier to swallowing or known swallowing disorder Diagnosis of severe developmental delay or mental retardation Significant brain pathology or seizure disorder that may affect oropharyngeal motor skills On medication with known effects on appetite or interactions with cyproheptadine

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Praveen Goday, MD, Principal Investigator — Medical College of Wisconsin Department of Pediatric Gastroenterology

REFERENCES:
- [Background] LAVENSTEIN AF, DACANEY EP, LASAGNA L, VANMETRE TE. Effect of cyproheptadine on asthmatic children. Study of appetite, weight gain, and linear growth. JAMA. 1962 Jun 16;180:912-6. doi: 10.1001/jama.1962.03050240008002. No abstract available. PMID 14462919
- [Background] Mahachoklertwattana P, Wanasuwankul S, Poomthavorn P, Choubtum L, Sriphrapradang A. Short-term cyproheptadine therapy in underweight children: effects on growth and serum insulin-like growth factor-I. J Pediatr Endocrinol Metab. 2009 May;22(5):425-32. doi: 10.1515/jpem.2009.22.5.425. PMID 19618661
- [Background] Sakata T, Ookuma K, Fukagawa K, Fujimoto K, Yoshimatsu H, Shiraishi T, Wada H. Blockade of the histamine H1-receptor in the rat ventromedial hypothalamus and feeding elicitation. Brain Res. 1988 Feb 16;441(1-2):403-7. doi: 10.1016/0006-8993(88)91423-0. PMID 3359243
- [Background] Homnick DN, Homnick BD, Reeves AJ, Marks JH, Pimentel RS, Bonnema SK. Cyproheptadine is an effective appetite stimulant in cystic fibrosis. Pediatr Pulmonol. 2004 Aug;38(2):129-34. doi: 10.1002/ppul.20043. PMID 15211696
- [Background] Homnick DN, Marks JH, Hare KL, Bonnema SK. Long-term trial of cyproheptadine as an appetite stimulant in cystic fibrosis. Pediatr Pulmonol. 2005 Sep;40(3):251-6. doi: 10.1002/ppul.20265. PMID 16015665
- [Background] Couluris M, Mayer JL, Freyer DR, Sandler E, Xu P, Krischer JP. The effect of cyproheptadine hydrochloride (periactin) and megestrol acetate (megace) on weight in children with cancer/treatment-related cachexia. J Pediatr Hematol Oncol. 2008 Nov;30(11):791-7. doi: 10.1097/MPH.0b013e3181864a5e. PMID 18989154
- [Background] Najib K, Moghtaderi M, Karamizadeh Z, Fallahzadeh E. Beneficial effect of cyproheptadine on body mass index in undernourished children: a randomized controlled trial. Iran J Pediatr. 2014 Dec;24(6):753-8. Epub 2014 Dec 12. PMID 26019782
- [Background] Sant'Anna AM, Hammes PS, Porporino M, Martel C, Zygmuntowicz C, Ramsay M. Use of cyproheptadine in young children with feeding difficulties and poor growth in a pediatric feeding program. J Pediatr Gastroenterol Nutr. 2014 Nov;59(5):674-8. doi: 10.1097/MPG.0000000000000467. PMID 24941960
- [Background] Powers SW, Byars KC, Mitchell MJ, Patton SR, Standiford DA, Dolan LM. Parent report of mealtime behavior and parenting stress in young children with type 1 diabetes and in healthy control subjects. Diabetes Care. 2002 Feb;25(2):313-8. doi: 10.2337/diacare.25.2.313. PMID 11815502

RESULTS

PARTICIPANT FLOW:
Groups:
- Continuous Cyproheptadine: Patients will receive standard of care behavior and nutritional interventions. They will receive cyproheptadine every day for a total of two months. Standard dose of 0.25 mg/kg divided BID will be used.
  Cyproheptadine
- Cycled Cyproheptadine: Patients will receive standard of care behavior and nutritional interventions. They will receive cyproheptadine every day for two weeks cycled with no cyproheptadine given for two weeks for a total of two months. Patients on cycled dosing will be given cyproheptadine for two weeks, then no medication for two weeks; repeating this cycle for the two month duration of study
  Cyproheptadine
Period: Overall Study
Arm/Group | No Cyproheptadine Treatment | Continuous Cyproheptadine | Cycled Cyproheptadine
Started | 2 | 2 | 0
Completed | 2 | 2 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: We had trouble recruiting patients for this study
Groups:
- Total: Total of all reporting groups
Arm/Group | No Cyproheptadine Treatment | Continuous Cyproheptadine | Cycled Cyproheptadine | Total
Number analyzed (Participants) | 2 | 2 | 0 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 4 (1.4) | 4 (1.4) |  | 4 (1.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 |  | 2
  Male | 1 | 1 |  | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 2 |  | 4

OUTCOME MEASURES:

1. Primary Outcome: Feeding Behavior Questionnaire
Description: Participants' guardians will complete the Mealtime Behavior Questionnaire (MBQ). This is a validated, 31-item, parent-report questionnaire assessing the mealtime behavior structure in young children above 2 years. The questionnaire measures variables including: 1) food refusals/avoidance; 2) food manipulation; 3) mealtime aggression and 4) choking/gagging/vomiting related to meals. Each behavior is assigned a frequency scale with 1 corresponding to "never" and 5 corresponding to "always." The MBQ then consist of a total score and four subcategory scores (listed above).
Time Frame: two months
Population: Too few patients to analyze
Arm/Group | No Cyproheptadine Treatment | Continuous Cyproheptadine | Cycled Cyproheptadine
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Anthropometrics: Skin Fold Thickness
Description: Change in skin fold thickness as measured by centimeters and z-score percentiles
Time Frame: two months
Population: Too few patients to analyze
Arm/Group | No Cyproheptadine Treatment | Continuous Cyproheptadine | Cycled Cyproheptadine
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Anthropometrics: Mid-arm Circumference
Description: Change in mid-arm circumference as measure by centimeters and z-score percentiles
Time Frame: two months
Population: Too few patients to be analyzed
Arm/Group | No Cyproheptadine Treatment | Continuous Cyproheptadine | Cycled Cyproheptadine
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Anthropometrics: BMI
Description: Change in BMI as measured by kilograms divided by meters squared and z-score percentiles
Time Frame: two months
Population: Too few patients to be analyzed
Arm/Group | No Cyproheptadine Treatment | Continuous Cyproheptadine | Cycled Cyproheptadine
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Anthropometrics: Height
Description: Change in height as measured in centimeters and z-score percentiles
Time Frame: two months
Population: Too few patients to be analyzed
Arm/Group | No Cyproheptadine Treatment | Continuous Cyproheptadine | Cycled Cyproheptadine
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Anthropometrics: Weight
Description: Change in weight as measured in kilograms and z-score percentiles
Time Frame: two months
Population: Too few patients to be analyzed
Arm/Group | No Cyproheptadine Treatment | Continuous Cyproheptadine | Cycled Cyproheptadine
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Percentage of Participants Experiencing Side Effects From Cyproheptadine
Description: Patients will answer affirmative or negative to a descriptive list of side effects commonly experienced when taking cyproheptadine. Examples of these descriptive variables include nausea, emesis, etc. Percentage of patients experiencing each side effect will be calculated and compared across the course of study.
Time Frame: two months
Population: Too few patients to be analyzed
Arm/Group | No Cyproheptadine Treatment | Continuous Cyproheptadine | Cycled Cyproheptadine
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: 24 Hour Diet Recall
Description: Change in calorie intake will be recorded
Time Frame: two months
Population: Too few patients to be analyzed
Arm/Group | No Cyproheptadine Treatment | Continuous Cyproheptadine | Cycled Cyproheptadine
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: Fatigue, Headache, Diarrhea, Vomiting, Constipation, Dry mouth, Nausea, sleepiness, Restlessness
Arm/Group | No Cyproheptadine Treatment | Continuous Cyproheptadine | Cycled Cyproheptadine
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/0
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/0

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed;

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes